CLINICAL TRIAL: NCT01540331
Title: Phase 4 Study to Evaluate Efficacy And Safety of Pneumatic Trabeculoplasty (PNT) in Subjects Affected by Primary Open Angle Glaucoma
Brief Title: Efficacy And Safety of Pneumatic Trabeculoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luigi Varano, MD, M. D., University of Catanzaro
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PNT01
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- PNT treatment (Experimental): all subjects enrolled in the study, that underwent PNT treatment
  Interventions: Device: "model 1000 PNT vacuum controller" (the vacuum device for ocular suction)

INTERVENTIONS:
Device: "model 1000 PNT vacuum controller" (the vacuum device for ocular suction) — A Pneumatic Trabeculoplasty treatment, composed of 3 single PNT applications at day 0, 7 and 90. Each treatment consist in a ocular pneumatic suction of 500inchHg administered for 60 seconds in perilimbal region through the device (model 1000 PNT vacuum controller). This suction is then repeated after a 5 minutes pause.
  Other Names: manifacturer: Ophthalmic International, Fountain Hills - AZ, USA

SUMMARY:
The purpose of this study is to evaluate prospectively the PNT safety and efficacy in term of IOP reduction in a group of previously or newly diagnosed glaucomatous subjects.

DETAILED DESCRIPTION:
A group of subjects affected by Primary Open Angle Glaucoma (POAG) underwent 3 PNT treatments to evaluate one-year efficacy in term of IOP reduction and one-year safety in term of incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Subjects affected by primary open angle glaucoma

Exclusion Criteria:

* Any local or systemic contraindication to timolol topical therapy
* Chronic iritis and/or uveitis in one or both eyes,
* History of inflammatory glaucoma,
* Hemorrhagic glaucoma,
* Post-traumatic glaucoma,
* Phacolytic glaucoma,
* Acute glaucomatocyclitic attack,
* Closed angle/narrow angle glaucoma in one or both eyes,
* Previous corneal transplantation,
* Proliferative diabetic retinopathy with/without iris neovascularisation,
* Significative disk cupping (90% of complete disk area),
* Large and severe perimetric defects (I. e. a central perimetric residual not above 10 central degrees),
* Dry/wet age related macular degeneration in one or both eyes,
* Previous glaucoma surgery (Laser therapy was not considered)
* Keratitis
* Severe dry eye disease,
* Corneal dystrophies
* High myopia (more than 6 dioptres)
* Peripheral retinal degenerations with risk of retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
intraocular pressure (IOP) | Patients will be followed for one year. Time-points:recruitment, Basal (30 days after recruitment), Follow-Up2 (30 days after basal), Follow-Up3 (3 months after basal), Follow-Up4 (6 months after basal), Follow-Up5 (one year after basal)
  to evaluate one-year intraocular pressure (IOP) reduction after a standard pneumatic trabeculoplasty (PNT) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Varano, M. D., Principal Investigator — University "Magna Graecia" of Catanzaro
Locations (1):
- University "Magna Graecia", Catanzaro, Italy